CLINICAL TRIAL: NCT04841564
Title: An Open Approach Versus Ultrasound Approach for Serratus Anterior Plane Block for Postoperative Analgesia After Modified Radical Mastectomy: A Non-inferiority Study
Brief Title: Open Versus Ultrasound Approach for Serratus Anterior Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Mahmoud Mohammed Alseoudy, Lecturer of anesthesia, ICU & pain management; Faculty of Medicine, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R.21.03.1262
Record Dates: First submitted 2021-04-07; First posted 2021-04-12 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Analgesia
Keywords: serratus anterior block; ultrasound; open; mastectomy
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ultrasound group (Active Comparator): serratus anterior plane block will be done through ultrasound guidance
  Interventions: Procedure: ultrasound approach of serratus anterior block
- Open group (Experimental): serratus anterior plane block will be done after mastectomy through the open wound
  Interventions: Procedure: open approach of serratus anterior block

INTERVENTIONS:
Procedure: ultrasound approach of serratus anterior block — After induction of general anesthesia, the ultrasound probe will be placed longitudinally oblique just below the mid-clavicle. After identifying the second rib, the probe will be moved caudally and laterally (obliquely), towards the mid-axillary line to identify the 3rd, 4th and 5th ribs.. The fascial plane between the serratus anterior muscle and latissimus dorsi muscle will be identified over the 4th rib in the mid-axillary region. The block will be performed with a needle (22-G, 50-mm) introduced in-plane to enter deep to the serratus anterior muscle, and 30 ml 0.25 bupivacaine will be injected.
  Other Names: ultrasound approach
  Arms: ultrasound group
Procedure: open approach of serratus anterior block — After resection of the breast and identification of the serratus anterior muscle, the surgeon will be asked to palpate the ribs below the clavicle and localize the fourth rib. A 22-G, 50-mm needle will be introduced deep to the serratus anterior muscle contacting the rib, and 30 ml 0.25 bupivacaine will be injected.
  Other Names: open approach
  Arms: Open group

SUMMARY:
Ultrasound-guided Serratus anterior plane (SAP) block is an interventional technique that recently gained popularity in the context of postoperative analgesia after breast surgery. Some limitations may be encountered during the use of ultrasound, such as obesity, tumor invasion of the surrounding muscles, which may lead to poor ultrasound image quality. The investigators hypothesized that an open approach to serratus anterior block by infiltration of local anesthetic between serratus anterior muscle and ribs after tumor excision during surgery would be non-inferior to ultrasound-guided approach where the primary endpoint of this prospective randomized blind controlled study will be the total dose of morphine consumed in the 1st postoperative 24 h. The patients will be randomly allocated to an open approach group and ultrasound approach group to serratus anterior block using computer-generated random numbers and sealed opaque envelops. For any statistical tests used results will be considered as statistically significant if P-value ≤0.05.

DETAILED DESCRIPTION:
Modified radical mastectomy (MRM) is one of the most common surgeries performed, and one that may be associated with significant acute postoperative pain in breast surgery. Acute postoperative pain is an independent risk factor in the development of chronic post-mastectomy pain.

Various regional anesthetic procedures have been tried to provide better acute pain control and, consequently, less chronic pain. They can reduce perioperative opiates requirement and thereby decreasing their possible side effects. These regional procedures include local wound infiltration, thoracic epidural, and thoracic paravertebral block (PVB). pectoral nerves block type-1 (PECSI), pectoral nerves block type-2 (PECS II), and serratus plane block.

Ultrasound-guided Serratus anterior plane (SAP) block is an interventional technique that recently gained popularity in the context of breast surgery. SAP block resulted in better hemodynamic stability, early ambulation, and reduced duration of hospitalization as well as hospital costs in postoperative breast patients.

Some limitations may be encountered during the use of ultrasound, such as obesity, tumor invasion of the surrounding muscles, which may lead to poor ultrasound image quality. Also, ultrasound use depends on equipment quality and investigator experience.

The investigators hypothesized that an open approach to serratus anterior block by infiltration of local anesthetic between serratus anterior muscle and ribs after tumor excision during surgery would be non-inferior to ultrasound-guided approach in providing analgesia to female patients undergoing modified radical mastectomy. The primary endpoint will be the total dose of morphine consumed in the 1st postoperative 24 h. secondary outcomes will be the time of the first analgesic request (duration of the pain-free periods after surgery in the1st postoperative 24 hours), postoperative visual analog score (VAS), postoperative modified Ramsay sedation score, and PONV (post-operative nausea and vomiting).

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) physical status scores of I and II
* Elective unilateral breast surgery (modified radical mastectomy)

Exclusion Criteria:

* Patient refusal to participate in the study.
* Allergy to any medications used in the study.
* Patients with coagulopathy
* patients with psychiatric disorders.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2021-04-10 (Actual); Primary Completion 2024-06-15 (Actual); Study Completion 2024-07-20 (Actual)

PRIMARY OUTCOMES:
Morphine consumption given as a rescue analgesia | Up to 24 hours after the procedure
  The amount of morphinel consumption in milligrams given as a rescue analgesia to patients when the vas score is more than 3

SECONDARY OUTCOMES:
The period for the first analgesic required | Up to 24 hours after the procedure
  duration of analgesia in minutes
Mean arterial blood pressure | Up to 24 hours after the procedure
  Mean arterial blood pressure in mmHg will be recorded at baseline before surgical incision and postoperatively at 1, 4, 8, 12, 24 hours
visual analogue score (VAS) at rest | Up to 24 hours after the procedure
  pain intensity will be assessed at rest with the 10 point visual analogue score (VAS) where 0 =no pain and 10 = the worst imaginable pain and the time points of measurements will be at 0, 1, 4, 8, 12 and 24 hours post-operatively.
postoperative complications | Up to 24 hours after the procedure
  Any postoperative events like nausea, vomiting, respiratory depression( respiratory rate less than 12), urine retention, pruritis, local anesthetic toxicity and pneumothorax will be recorded.
Heart rate | Up to 24 hours after the procedure
  Heart rate in beats per minute will be recorded at baseline before surgical incision and postoperatively at 1, 4, 8, 12, 24 hours
visual analogue score (VAS) at shoulder movement | Up to 24 hours after the procedure
  pain intensity will be assessed at shoulder movement with the 10 point visual analogue score (VAS) where 0 =no pain and 10 = the worst imaginable pain and the time points of measurements will be at 0, 1, 4, 8, 12 and 24 hours post-operatively.

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud M Alseoudy, MD, Principal Investigator — mansoura university, faculty of medicine
Locations (1):
- Department of Anesthesia, Mansoura University Hospitals, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mohammed ALseoudy M, Abd El-Ghaffar Saleh M, Saleh Elbalka S, Elmetwally Farahat T, Abdellatif Elebedy D, Elsayed Ahmed S. An open approach versus ultrasound approach for deep serratus anterior plane block for postoperative analgesia after modified radical mastectomy: A randomized controlled trial. Rev Esp Anestesiol Reanim (Engl Ed). 2025 Nov;72(9):501902. doi: 10.1016/j.redare.2025.501902. Epub 2025 Sep 4. PMID 40914287